CLINICAL TRIAL: NCT07092371
Title: Smartphone Multimodal Health Intervention for Neurological Enhancement (SHINE) in High Stroke-risk Population: a Randomized Trial
Brief Title: Smartphone Multimodal Health Intervention for Neurological Enhancement (SHINE)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SHINE
Record Dates: First submitted 2025-05-12; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-05

CONDITIONS: Cognitive Impairment; Dementia; Artificial Intelligence (AI); Stroke; Cognitive Decline
Keywords: stoke; cognitive impairment; cognitive decline; dementia; Artificial intelligence (AI)
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Multimodal Intervention Group (Active Comparator): Participants will receive a 6-month multimodal intervention through a digital platform, including: (1) Personalized cognitive training; (2) Self-monitoring and management of stroke risk factors including hypertension, dyslipidemia, diabetes, smoking and obesity; (3) Smart wristband-based exercise monitoring and management; (4) Smart wristband-based sleep monitoring and management; (5) Health dietary recording and guidance
  Interventions: Behavioral: Digital Multimodal Intervention
- Standard health counseling (No Intervention): standard educational materials and care at baseline

INTERVENTIONS:
Behavioral: Digital Multimodal Intervention — Participants will undergo a 6-month multimodal intervention via a digital platform, which includes: (1) Personalized cognitive training; (2) Self-monitoring and management of stroke risk factors including hypertension, dyslipidemia, diabetes, smoking and obesity; (3) Smart wristband-based exercise monitoring and management; (4) Smart wristband-based sleep monitoring and management; (5) Health dietary recording and guidance
  Arms: Digital Multimodal Intervention Group

SUMMARY:
This randomized controlled trial will enroll individuals aged ≥ 40 years without dementia who are at high risk for stroke, collecting multi-modal MRI imaging, serum, and fecal samples to investigate the effects of a smartphone-based multimodal health intervention on cognitive function measured using digital-evaluated cognitive scores.

DETAILED DESCRIPTION:
The Smartphone-based multimodal Health Intervention for Neurological Enhancement (SHINE) trial is designed to test the impact of a 6-month artificial intelligence(AI)-assisted intervention utilizing smartphone-based multimodal lifestyle and stroke risk factor management on 1036 participants aged 40 years and above who are without dementia and are at high risk for stroke. The multimodal digital program integrated adaptive cognitive training, personalized cardiovascular risk management, smart wristband-based physical activity and sleep monitoring, and dietary guidance, all delivered through a smartphone application incorporating behavioral change and AI techniques. Participants in the intervention group will receive the lifestyle and stroke risk factors management, while participants in the control group will receive standard educational materials and care. The investigation will explore potential mediators and modifiers of the intervention's effects by collecting various cardiovascular risk factors, serum samples, fecal samples, neuropsychological assessment results, and multi-modal magnetic resonance imaging at baseline, 6 months, 1 year, and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 40 years
* High risk of stroke (with ≥ 3 of 8 stroke risk factors, including hypertension, dyslipidemia, diabetes, atrial fibrillation or valvular heart disease, smoking history, obvious overweight or obesity, lack of exercise, family history of stroke, or with transient ischemic attack)
* Written informed consent available
* Primary school education or above
* Proficient in using smartphones
* Willingness to complete all assessments and participate in follow-up

Exclusion Criteria:

* previously diagnosed dementia
* Suspected dementia after clinical assessment by study physician at screening visit
* Previous history of major head trauma and any intracranial surgery
* Intracranial abnormalities, such as intracerebral hemorrhage, subarachnoid hemorrhage and other space occupying lesions
* Extrapyramidal symptoms or mental illness which may affect neuropsychological measurement
* Severe loss of vision, hearing, or communicative ability
* Patients presenting a malignant disease with life expectancy < 3 years
* Participation in an ongoing investigational drug study

Exit Criteria:

* Not meet the inclusion criteria
* For any poor adherence, not comply with the requirements of the follow-up, or safety reasons determined by investigator
* Any adverse or serious adverse events during the study period judged by Investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1036 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Global cognitive function change assessed with Z-score of a digital cognitive assessment protocol | 6 months
  Primary Outcome

SECONDARY OUTCOMES:
Cognitive function change assessed by Montreal Cognitive Assessment (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 6 months, 1 year, 2 years
  Secondary Outcome
Cognitive function change assessed with Mini-Mental State Examination (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 6 months, 1 year, 2 years
  Secondary Outcome
Metabolite composition to measure the metabolite profiles in participants' faecal samples and serum samples | 6 months, 1 year, 2 years
  Secondary Outcome
The Oriental Intervention for Enhanced Neurocognitive health (ORIENT) diet score (minimum value = 0, maximum value = 14, and higher scores mean a better outcome) | 6 months, 1 year, 2 years
  Secondary Outcome
Sleep quality assessed by Pittsburgh sleep quality index (minimum value = 0, maximum value = 21, and higher scores mean a worse outcome) | 6 months, 1 year, 2 years
  Secondary Outcome
Dementia and cerebrovascular events incidence | 2 years, 5 years
  Secondary Outcome
Gut microbiota determined by measuring specific bacterial levels in the fecal samples | 6 months, 1 year, 2 years
  Secondary Outcome
Frequency of digital platform usage for lifestyle and risk factor management (number of weekly platform feature accesses, tracked through platform analytics) | 6 months, 1 year, 2 years
  Secondary Outcome
Completeness of data uploads on digital platform | 6 months, 1 year, 2 years
  Secondary Outcome
Change in waist circumference if overweight/obese | 6 months, 1 year, 2 years
  Secondary Outcome
Change in body mass index (BMI) if overweight/obese | 6 months, 1 year, 2 years
  Secondary Outcome
working memory domain cognitive score change assessed with a digital cognitive assessment protocol (higher scores mean a better outcome) | 6 months, 1 year, 2 years
  Secondary Outcome
executive function domain cognitive score change assessed with a digital cognitive assessment protocol (higher scores mean a better outcome) | 6 months, 1 year, 2 years
  Secondary Outcome
language domain cognitive score change assessed with a digital cognitive assessment protocol (higher scores mean a better outcome) | 6 months, 1 year, 2 years
  Secondary Outcome
visual motor speed domain cognitive score change assessed with a digital cognitive assessment protocol (higher scores mean a better outcome) | 6 months, 1 year, 2 years
  Secondary Outcome
visual spatial function domain cognitive score change assessed with a digital cognitive assessment protocol (higher scores mean a better outcome) | 6 months, 1 year, 2 years
  Secondary Outcome
memory and recognition domain cognitive score change assessed with a digital cognitive assessment protocol (higher scores mean a better outcome) | 6 months, 1 year, 2 years
  Secondary Outcome
Visual Analogue Scale (VAS) score of EuroQol Five Dimension Five Level (EQ-5D-5L) Questionnaire (higher VAS score indicates better health status) | 6 months, 1 year, 2 years
  Secondary Outcome
Utility index of EuroQol Five Dimension Five Level (EQ-5D-5L) Questionnaire (higher utility index indicates better health-related quality of life) | 6 months, 1 year, 2 years
  Secondary Outcome
Change in level of physical activity assessed with daily step count | 6 months, 1 year, 2 years
  Secondary Outcome
Change in level of physical activity assessed with Metabolic Equivalent of Task [MET] per week, higher MET per week means higher physical activity levels | 6 months, 1 year, 2 years
  Secondary Outcome
Change in systolic blood pressure (SBP) in participants with self-report history of hypertension | 6 months, 1 year, 2 years
  Secondary Outcome
Change in diastolic blood pressure (DBP) in participants with self-report history of hypertension | 6 months, 1 year, 2 years
  Secondary Outcome
Change in fasting blood glucose levels in participants with self-report history of hypertension in participants with self-report history of diabetes | 6 months, 1 year, 2 years
  Secondary Outcome
Change in insulin resistance assessed by Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) in participants with self-report history of diabetes (higher HOMA-IR indicatehigher insulin resistance) | 6 months, 1 year, 2 years
  Secondary Outcome
Change in glycated hemoglobin (HbA1c) levels (%) in participants with self-report history of diabetes | 6 months, 1 year, 2 years
  Secondary Outcome
Change in low-density lipoprotein cholesterol (LDL-C) levels in participants with self-report history of dyslipidemia | 6 months, 1 year, 2 years
  Secondary Outcome
Change in high-density lipoprotein cholesterol (HDL-C) levels in participants with self-report history of dyslipidemia | 6 months, 1 year, 2 years
  Secondary Outcome
Change in total cholesterol (TC) levels in participants with self-report history of dyslipidemia | 6 months, 1 year, 2 years
  Secondary Outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affilated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No